CLINICAL TRIAL: NCT01517282
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib Study to Evaluate the Safety and Pharmacokinetics of MOR103, a Human Antibody to GM-CSF, in Patients With Multiple Sclerosis
Brief Title: Phase Ib Study to Evaluate MOR103 in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-001064-22
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Otilimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MOR103 0.5 mg/kg (Experimental): 6 doses of MOR103 0.5 mg/kg administered on Days 1 (Baseline), 15 (Visit 2), 29 (Visit 3), 43 (Visit 4), 57 (Visit 5), and 71 (Visit 6).
  Interventions: Biological: MOR103
- MOR103 1.0 mg/kg (Experimental): 6 doses of MOR103 1.0 mg/kg administered on Days 1 (Baseline), 15 (Visit 2), 29 (Visit 3), 43 (Visit 4), 57 (Visit 5), and 71 (Visit 6).
  Interventions: Biological: MOR103
- MOR103 2.0 mg/kg (Experimental): 6 doses of MOR103 2.0 mg/kg administered on Days 1 (Baseline), 15 (Visit 2), 29 (Visit 3), 43 (Visit 4), 57 (Visit 5), and 71 (Visit 6).
  Interventions: Biological: MOR103
- Placebo (Placebo Comparator): 6 doses of placebo administered on Days 1 (Baseline), 15 (Visit 2), 29 (Visit 3), 43 (Visit 4), 57 (Visit 5), and 71 (Visit 6).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MOR103 — Anti-GM-CSF monoclonal antibody
  Arms: MOR103 0.5 mg/kg; MOR103 1.0 mg/kg; MOR103 2.0 mg/kg
Other: Placebo — Placebo to anti-GM-CSF monoclonal antibody
  Arms: Placebo

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease associated with central nervous system (CNS) demyelination and subsequent axonal degeneration. Multiple sclerosis exhibits an unpredictable and variable clinical course.

Multiple sclerosis plaques contain numerous types of cells and infiltrating macrophages have been identified to contribute significantly to demyelination in both clinical MS and animal models of MS. Granulocyte-macrophage colony-stimulating factor (GM CSF) stimulates proliferation and activation of macrophages, monocytes, neutrophils, eosinophils, dendritic cells and microglia with subsequent induction of proinflammatory biomolecules.

Therefore blocking GM CSF activity might be a therapeutic approach for the treatment of MS.

DETAILED DESCRIPTION:
Recent clinical studies demonstrated a possible dysregulation of the balance of pro and anti inflammatory lymphocytes, which may contribute to the pathogenesis of MS.

It was shown in animal models of EAE that during the disease effect or phase GM CSF sustained neuroinflammation via myeloid cells that infiltrate the CNS proving an essential role of GM CSF in encephalitogenicity.

ELIGIBILITY:
Key Inclusion Criteria:

Outpatients with a diagnosis of RRMS or SPMS, who are currently not being treated and who have at least 1 of the following:

* At least 1 documented relapse within 1 year before Screening, or
* Two documented relapses within the past 2 years before Screening, or
* A new gadolinium (Gd)-enhancing lesion on magnetic resonance imaging (MRI) T1-weighted imaging within 1 year before Screening, or
* A new T2 lesion on MRI within 1 year before Screening. The patient must have 10 or less, Gd-enhancing lesions per T1-weighted MRI at Screening as assessed by a central reader.

The patient must be able and willing to ambulate, with an Expanded Disability Status Scale (EDSS) score of ≥ 2.0 and ≤ 6.5 at both the Screening Visit and the Baseline Visit

Key Exclusion Criteria:

1. A patient with primary progressive MS (PPMS)
2. A patient who has previously received at any time any of the following

   * B-cell or T-cell depleting therapies
   * Cytotoxic agents, any immunosuppressive/immunomodulating agents
3. A patient who has not stabilized, in the opinion of the investigator
4. A patient with any medical condition or uncontrolled disease states other than MS requiring or likely to require systemic treatment with corticosteroids or other immune compromising agents
5. A patient with current or a history of major chronic inflammatory autoimmune diseases other than MS
6. A patient with any type of infection
7. Patients on chronic prophylactic or suppressive antibiotic, antifungal,or antiviral agents
8. A patient with a history of tuberculosis.
9. A patient with any signs of excretory hepatic or kidney dysfunction
10. A patient with a positive test for Hepatitis B or Hepatitis C

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman P Korolkiewicz, MD, PhD, Study Director — MorphoSys AG
Locations (5):
- Morphosys Investigative Site, Berlin, Germany
- Poland (2):
  - Morphosys Investigative Site, Gdansk
  - Morphosys Investigative Site, Poznan
- United Kingdom (2):
  - Morhosys Investigative Site, Manchester
  - MorphoSys Investigative Site, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and screened between 2 January 2012 and 22 July 2013 at 5 trial centers in Europe (1 in Germany, 2 in Poland, and 2 in the United Kingdom). Screening could occur between 10 and 35 days prior to dosing on day 1. Subject eligibility was determined at the screening visit and confirmed before the first dose on day 1.
Groups:
- MOR103 0.5 mg/kg: MOR103 0.5 mg/kg administered intravenously every 2 weeks for a total of 6 doses.
- MOR103 1.0 mg/kg: MOR103 1.0 mg/kg administered intravenously every 2 weeks for a total of 6 doses.
- MOR103 2.0 mg/kg: MOR103 2.0 mg/kg administered intravenously every 2 weeks for a total of 6 doses.
- Pooled Placebo: Placebo administered intravenously once every 2 weeks for a total of 6 doses
Period: Overall Study
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Started | 9 (One patient was randomized but did not receive study medication based on the investigator's decision) | 8 | 9 (1 patient completed the trial, but received only 4 doses of medication and 2 MRIs due to pregnancy) | 6
Completed | 8 | 7 | 8 | 5
Not Completed | 1 | 1 | 1 | 1
Not completed — Consent withdrawn | 0 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received 1 or more dose of placebo or MOR103 (safety population).
Groups:
- Total: Total of all reporting groups
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo | Total
Number analyzed (Participants) | 8 | 8 | 9 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.63) | 48.6 (4.98) | 48.3 (11.47) | 43.5 (15.03) | 47.3 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 3 | 20
  Male | 4 | 2 | 2 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 7 | 8 | 9 | 5 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 2 | 1 | 1 | 2 | 6
  Germany | 2 | 5 | 3 | 2 | 12
  United Kingdom | 4 | 2 | 5 | 2 | 13
Diagnosis [Number; unit: participants]
  Relapsing-remitting multiple sclerosis | 7 | 6 | 6 | 6 | 25
  Secondary progressive multiple sclerosis | 1 | 1 | 3 | 0 | 5
  Unknown | 0 | 1 | 0 | 0 | 1
Time since diagnosis [Mean (Standard Deviation); unit: years] | 5.6 (8.68) | 13.1 (7.38) | 10.7 (8.97) | 5.5 (7.66) | 9.0 (8.51)
Gadolinium (Gd)-enhancing lesions [Number; unit: participants]
  1 or more Gd-enhancing lesions | 3 | 3 | 1 | 3 | 10
  No Gd-enhancing lesions | 5 | 5 | 8 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Patients With Treatment-emergent Adverse Events (TEAEs) or Treatment-emergent Serious Adverse Events (TESAEs)
Description: The safety of multiple doses of MOR103 in patients with relapsing-remitting or secondary progressive multiple sclerosis (MS) was assessed by evaluation of the incidence of TEAEs and TESAEs. A full listing of adverse events recorded during this trial can be found in the Adverse Events section. AEs were regarded as treatment emergent if they started on or after the first date of study drug administration or if they were present prior to the first date of study drug administration and increased in severity or relationship to study drug during the study. AEs were coded using MedDRA version 16.1
Time Frame: From the first dose (week 0) to study endpoint (week 20)
Population: All subjects who received 1 or more dose of placebo or MOR103 (safety population).
Measure: Number; unit: percentage of participants
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 6
percentage of participants
  Any TEAE | 100 | 100 | 88.9 | 100
  Any TEAE related to treatment | 75.0 | 50.0 | 33.3 | 83.3
  Any TEAE with MS exacerbation/relapse | 62.5 | 12.5 | 0.0 | 50.0
  Any TESAE | 0 | 12.5 | 0 | 16.7

2. Secondary Outcome: Percentages of Patients Negative for Anti-MOR103 Antibodies in Serum Samples
Description: To assess the potential immunogenicity of MOR103, a central bioanalytical laboratory (Eurofins Medinet BV, Breda, The Netherlands) tested serum samples obtained at baseline and at 3 post-treatment time points (week 14, week 16, and week 20/end of study) for anti-MOR103 antibodies.
Time Frame: Baseline, week 14, week 16, and week 20/end of study
Population: All subjects who received 1 or more dose of placebo or MOR103 (safety population). Data were missing for 1 patient each in the MOR103 1.0 mg/kg and 2.0 mg/kg groups at week 14 and week 16. Data were also missing for 1 patient in the placebo group at all post-baseline timepoints (week 14, 16, and 20).
Measure: Number; unit: percentage of participants
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 6
percentage of participants
  Baseline | 100 | 100 | 100 | 100
  Week 14 | 100 | 100 | 100 | 100
  Week 16 | 100 | 100 | 100 | 100
  Week 20 | 100 | 100 | 100 | 100

3. Secondary Outcome: Mean Serum Concentration of MOR103 Over Time
Description: MOR103 serum levels were measured at each visit. At all visits during the dosing period (weeks 0, 2, 6, 8, and 10), serum samples were taken before MOR103 administration (pre-dose) and 1 hour after the dose. In addition, at week 0 (first dose) and week 10 (last dose), additional samples were obtained at 2 hours and 4 hours after MOR103 administration. At visits that followed the dosing period (weeks 12, 14, 16, and 20), a single serum sample was obtained at any time during the visit.
Time Frame: Week 0 (dose 1) to week 20 (end of study)
Population: Pharmacokinetic (PK) analyses were conducted on the PK set, which included all MOR103-treated patients except for 2 patients who discontinued after 2 doses of trial medication (one each in the 1.0 and 2.0 mg/kg groups). PK data were not available for all patients at each time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg
Number analyzed (Participants) | 8 | 7 | 8
mg/L
  Week 0: Pre-dose | 0 (0) | 3.778 (9.995) | 0 (0)
  Week 0: 1 hour after 1st dose | 7.686 (3.00) | 17.907 (3.180) | 34.834 (6.770)
  Week 0: 2 hours after 1st dose | 7.935 (1.827) | 17.715 (3.004) | 33.600 (6.336)
  Week 0: 4 hours after 1st dose | 7.458 (1.337) | 16.765 (2.816) | 30.259 (4.921)
  Week 2: Pre-dose | 0.555 (0.225) | 1.422 (0.588) | 2.372 (0.779)
  Week 2: 1 hour after 2nd dose | 8.053 (0.839) | 22.021 (6.700) | 39.536 (7.535)
  Week 4: Pre-dose | 1.671 (2.547) | 1.544 (0.283) | 3.070 (1.205)
  Week 4: 1 hour after 3rd dose | 6.972 (2.947) | 21.351 (5.435) | 37.605 (5.734)
  Week 6: Pre-dose | 0.924 (0.322) | 1.831 (0.297) | 3.494 (1.440)
  Week 6: 1 hour after 4th dose | 9.298 (1.155) | 21.836 (6.077) | 42.200 (15.467)
  Week 8: Pre-dose | 0.934 (0.386) | 2.138 (0.867) | 3.654 (1.539)
  Week 8: 1 hour after 5th dose | 9.120 (1.618) | 22.283 (4.738) | 40.464 (4.432)
  Week 10: Pre-dose | 0.929 (0.323) | 2.143 (0.884) | 3.584 (1.859)
  Week 10: 1 hour after 6th and last dose | 8.536 (1.787) | 23.675 (7.695) | 38.853 (6.720)
  Week 10: 2 hours after 6th and last dose | 8.820 (2.037) | 21.204 (6.972) | 37.361 (8.238)
  Week 10: 4 hours after 6th and last dose | 7.942 (1.105) | 20.960 (6.521) | 35.652 (6.106)
  Week 12 | 0.907 (0.240) | 2.065 (0.606) | 3.966 (2.069)
  Week 14 | 0.351 (0.140) | 0.869 (0.341) | 1.318 (0.419)
  Week 16 | 0.175 (0.072) | 0.416 (0.205) | 0.720 (0.480)
  Week 20 | 0.118 (0.076) | 0.179 (0.097) | 0.118 (0.034)

4. Secondary Outcome: Mean Maximum MOR103 Concentration (Cmax) After the First and Last MOR103 Doses
Description: At the week 0 (first dose) and week 10 (last dose) visits, serum samples were obtained at pre-dose and at 1, 2, and 4 hours after the dose. Cmax values for each patient were calculated based on these data, and the mean Cmax values for the dose cohort are presented here. Because Cmax refers to the maximum serum concentration, only one value is presented for each dose cohort on each day; values at each PK time point are not applicable, as they represent the concentration of MOR103, but not the Cmax.
Time Frame: Week 0 (first dose) and week 10 (last dose)
Population: Pharmocokinetic (PK) analyses were conducted on the PK set, which included all MOR103-treated patients except for 2 patients who discontinued after 2 doses of trial medication (one each in the 1.0 and 2.0 mg/kg groups). PK data for the last dose were missing for one patient in the MOR103 2.0 mg/kg group (n = 7).
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg
Number analyzed (Participants) | 8 | 7 | 8
mg/L
  Week 0 (first dose) | 8.60 (2.08) | 18.70 (2.97) | 35.67 (6.73)
  Week 10 (last dose) | 9.03 (1.81) | 22.53 (7.71) | 40.37 (6.37)

5. Secondary Outcome: Mean Time to Maximum MOR103 Concentration (Tmax) After the First and Last MOR103 Doses
Description: At the week 0 (first dose) and week 10 (last dose) visits, serum samples were obtained at pre-dose and at 1, 2, and 4 hours after the dose. Tmax values for each patient were calculated based on these data, and the mean Tmax values for the dose cohort are presented here. Because Tmax refers to the time to maximum serum concentration, only one value is presented for each dose cohort on each day; values at each PK time point are not applicable.
Time Frame: Week 0 (first dose) and week 10 (last dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg
Number analyzed (Participants) | 8 | 7 | 8
hour
  Week 0 (first dose) | 1.89 (1.01) | 1.49 (1.12) | 1.39 (0.50)
  Week 10 (last dose) | 2.03 (0.89) | 1.44 (1.13) | 1.31 (0.47)

6. Secondary Outcome: Accumulation Ratio for Area Under the MOR103 Serum Concentration Versus Time Curve (AUC) Over One Dosing Interval: Ratio of Week 10 (Last Dose) AUC to Week 0 (First Dose) AUC
Description: At week 0 (first dose) and week 10 (last dose), serum samples were obtained at pre-dose and at 1, 2, 4, and 336 hours after start of dosing. To calculate the accumulation ratio, the apparent AUC calculated for the last dose was divided by the apparent AUC following the first dose using the described time points for each dosing. Because AUC is a summary outcome, only one value is presented for each dose cohort on each day; values at each PK time point are not applicable.
Time Frame: Week 0 (first dose) and week 10 (last dose)
Population: Pharmocokinetic (PK) analyses were conducted on the PK set, which included all MOR103-treated patients except for 2 patients who discontinued after 2 doses of trial medication (one each in the 1.0 and 2.0 mg/kg groups). Data were missing for one patient in the MOR103 2.0 mg/kg group (n = 7).
Measure: Mean (Standard Deviation); unit: ratio of AUC values
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg
Number analyzed (Participants) | 8 | 7 | 7
ratio of AUC values | 1.20 (0.13) | 1.31 (0.20) | 1.32 (0.22)

7. Secondary Outcome: Number of New T1 Gadolinium-enhancing Lesions
Description: Magnetic resonance imaging (MRI) tests were performed at screening (to confirm subject eligibility) and at Weeks 4, 8, 2, and 16. MRIs at post-screening time points were used to assess the number of new lesions as revealed by gadolinium (Gd) enhancement. Gd-enhanced MRIs reveal new brain lesions reflecting areas of active inflammation. MRI images were assessed centrally by Synarc A/S (Hamburg, Germany).
Time Frame: Week 4, week 8, week 12, and week 16.
Population: MRIs were performed in the safety population (all patients who received at least 1 dose of MOR103 or placebo). However, MRIs at Weeks 12 and 16 were not mandatory per protocol. The number of patients evaluated at Weeks 4, 8, 12, and 16 were:
  MOR103 0.5 mg/kg: 8,8,8,8 MOR103 1.0 m/kg: 6,6,6,6 MOR103 2.0 mg/kg: 8,7,7,7 Placebo: 6, 6, 4, 5
Measure: Number; unit: Number of new T1 Gd-enhancing lesions
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 6
Number of new T1 Gd-enhancing lesions
  Week 4 | 8 | 1 | 1 | 4
  Week 8 | 3 | 2 | 1 | 3
  Week 12 | 11 | 3 | 1 | 0
  Week 16 | 8 | 6 | 1 | 3

8. Secondary Outcome: Number of New or Enlarging T2 Lesions
Description: T2-weighted magnetic resonance imaging (MRI) tests were performed at Weeks 8, 12, and 16 to assess the number of new or enlarging T2 brain lesions, a sign of MS activity. MRI images were assessed centrally by Synarc A/S (Hamburg, Germany).
Time Frame: Week 8, week 12, and week 16.
Population: MRIs were performed in the safety population (all patients who received at least 1 dose of MOR103 or placebo). However, MRIs at Weeks 12 and 16 were not mandatory per protocol. The number of patients evaluated at Weeks 8, 12, and 16 were:
  MOR103 0.5 mg/kg: 8,8,8 MOR103 1.0 m/kg: 6,6,6 MOR103 2.0 mg/kg: 7,7,7 Placebo: 6, 4, 5
Measure: Number; unit: Number of new or enlarging T2 lesions
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 6
Number of new or enlarging T2 lesions
  Week 8 | 23 | 3 | 2 | 9
  Week 12 | 9 | 3 | 0 | 1
  Week 16 | 16 | 9 | 0 | 5

ADVERSE EVENTS:
Time Frame: From first dose of study medication to last visit (week 20)
Description: Patients were examined for adverse events (AEs) at all study visits. Data for treatment-emergent AEs (AEs occurring or worsening after the first dose of medication) are presented here.
Arm/Group | MOR103 0.5 mg/kg | MOR103 1.0 mg/kg | MOR103 2.0 mg/kg | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOR103 0.5 mg/kg (N=8) | MOR103 1.0 mg/kg (N=8) | MOR103 2.0 mg/kg (N=9) | Pooled Placebo (N=6)
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOR103 0.5 mg/kg (N=8) | MOR103 1.0 mg/kg (N=8) | MOR103 2.0 mg/kg (N=9) | Pooled Placebo (N=6)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 3 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 2
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Influenza-like illness (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 1 | 4
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 0 | 0
Hemoglobin urine present (Investigations) | 0 | 0 | 1 | 0
Hysteroscopy (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 | 0 | 0 | 0
Peak expiratory flow rate decreased (Investigations) | 1 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 4 | 1 | 0 | 3
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 3 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intra-uterine contraceptive device (Surgical and medical procedures) | 0 | 0 | 0 | 1
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Key limitations of this trial include its small sample size and limited duration. Efficacy assessments were not made in this study. Larger clinical trials will be required to evaluate the potential of MOR103 in treating patients with MS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information supplied by MorphoSys is considered confidential until publication and shall not be disclosed without prior written consent from MorphoSys. No data can be published in any format without prior approval of MorphoSys, which has final decision on approving submissions for publication. In the event of disagreement in the content of a publication, both the Author's and MorphoSys' opinion will be fairly and sufficiently represented in the publication.